CLINICAL TRIAL: NCT00269906
Title: Chimeric Anti-Platelet Therapy (Abciximab) in Unstable Angina Refractory to Standard Medical Therapy Trial (CAPTURE)
Brief Title: A Study Evaluating the Efficacy and Safety of Abciximab, an Anti-Platelet Therapy, in Patients With Unstable Angina Not Responding to Standard Medical Therapy Who Are Eligible for Coronary Angioplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006271
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Angina, Unstable; Angioplasty, Transluminal, Percutaneous Coronary
Keywords: Angina, unstable; Angioplasty, transluminal, percutaneous coronary; Abciximab
MeSH Terms: conditions — Angina, Unstable | interventions — Abciximab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Abciximab (c7E3 Fab) (Experimental): Participants will receive 0.25 milligram per kilogram (mg/kg) of body weight abciximab as bolus intravenous injection followed by continuous infusion of abciximab at rate of 10 microgram per minute for at least 18 hours but not longer than 26 hours.
  Interventions: Drug: Abciximab
- Placebo (Placebo Comparator): Participants will receive matching placebo as bolus IV injection followed by continuous infusion of matching placebo for at least 18 hours but no longer than 26 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Abciximab
  Other Names: c7E3 Fab
  Arms: Abciximab (c7E3 Fab)
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of abciximab, an anti-platelet therapy, versus placebo in patients with unstable angina who are not responding to standard medical therapy and who are eligible for coronary angioplasty.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled study to evaluate the safety and efficacy of abciximab, an anti-platelet therapy, in patients with unstable angina who are not responding to standard medical therapy and who are eligible for coronary angioplasty. The primary outcomes of the study include any of the following within 30 days: the number of deaths from any cause, myocardial infarctions or the number of recurrent ischemic events requiring urgent intervention (such as a coronary artery bypass surgery, repeat coronary angioplasty, coronary stent placement, or intra-aortic balloon pump). Please see attached results.

Patients will be treated with abciximab or matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory angina as evidenced by at least one episode of ischemia (chest pain and/or ST-T changes) despite bed rest and at least 2 hours of treatment with oral or intravenous nitrates and intravenous heparin, or persistent newly developed negative T-waves occurring or continuing after at least 2 hours of treatment with oral or intravenous nitrates and intravenous heparin
* Having clinical signs and symptoms of angina at rest or minimal exertion with dynamic ST-segment and/or T-wave changes
* Having an episode of chest pain within 48 hours prior to the start of study agent administration
* Having a culprit lesion in a single native coronary vessel suitable for angioplasty on the qualifying angiogram

Exclusion Criteria:

* Patients who have had a recent myocardial infarction, unless CK has returned to less than twice the upper limit of normal
* Having features of ongoing ischemia that would require immediate intervention, or had a percutaneous transluminal coronary angioplasty (PTCA) within the past 24 hours
* Having an unprotected occlusion of the main left coronary artery > 50%, a culprit lesion located in a venous or arterial bypass graft, or recent bleeding or a condition associated with increased bleeding risk
* Receiving concurrent administration of oral anticoagulants at the time of study entry, administration of intravenous dextran (prior to or planned for use during angioplasty), or planned administration of thrombolytic agent prior to or during angioplasty
* Having persistent hypertension at admission despite treatment, or a platelet count less than 100,000 per millimeter cubed

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1265 (Actual)
Dates: Start 1993-05; Primary Completion 1995-12 (Actual); Study Completion 1995-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants who Died From Any Cause | Up to 30 Days
Number of Participant with any one of these: Myocardial Infraction, Recurrent Ischemic Events Requiring Urgent Intervention (Coronary Artery Bypass Surgery, Repeat Coronary Angioplasty, Coronary Stent Placement, Intra-aortic Balloon Pump) | Up to 30 Days

SECONDARY OUTCOMES:
Number of Participants With New Ischemia | From onset of infusion to percutaneous transluminal coronary angioplasty (PTCA), and from PTCA through 24 hours after PTCA
Number of Participants With PTCA Complications | From onset of infusion to PTCA, and from PTCA through 24 hours after PTCA
Number of Participants With use of Thrombolytic Agents in the Catheterization | Day 1
Number of Participants With use of a Balloon Perfusion Catheter During Procedure | Day 1
Number of Particpants With Late Major Clinical Events | From Day 30 up to 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Result] Randomised placebo-controlled trial of abciximab before and during coronary intervention in refractory unstable angina: the CAPTURE Study. Lancet. 1997 May 17;349(9063):1429-35. PMID 9164316